CLINICAL TRIAL: NCT07337512
Title: Moringa Oleifera and Phoenix Dactylifera L. Effects on Cortisol and Breast Milk in Postpartum Depression: A Randomized Controlled Trial
Brief Title: Moringa Oleifera and Phoenix Dactylifera L. Effects on Cortisol and Breast Milk in Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melania Asi (Other)
Collaborators: Indonesia-MoH (Other Government)
Responsible Party: Sponsor-Investigator, Melania Asi, Director, Health Polytechnic, Ministry of Health, Kendari
Organization: Health Polytechnic, Ministry of Health, Kendari (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DP.04.03/F.XXXVI.15/010/2024; 7011.PKPT.001.43321 (Other Grant/Funding Number: Ministry of health, indonesia)
Record Dates: First submitted 2025-12-06; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Depression (PPD)
Keywords: Moringa oleifera Leaf; Phoenix dactylifera L; Salivary Cortisol; Breast Milk; Postpartum Mother; Depression
MeSH Terms: conditions — Depression, Postpartum; Depression | interventions — flocculant protein MO 2.1, Moringa oleifera

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3 (Active Comparator): This study employed a three-arm design over 28 days comparing two active interventions against placebo control. The Phoenix dactylifera L. group received 120g daily dates (40g portions thrice daily) using food-grade certified products with precise digital scaling (±0.1g accuracy) and controlled storage in airtight containers with humidity regulation. The Moringa oleifera group received pharmaceutical-grade capsules at 1000mg daily (500mg twice daily) with analytical balance verification (±0.1mg) and amber glass storage for light protection. The placebo group maintained regular three-daily meals without additional intervention. Both active groups utilized standardized measurement protocols, quality-certified materials, and comprehensive documentation systems including food diaries and visual monitoring to ensure intervention fidelity and participant compliance throughout the study period.
  Interventions: Drug: Phoenix dactylifera L; Drug: Moringa oleifera; Other: Placebo: consumed food three times a day

INTERVENTIONS:
Drug: Phoenix dactylifera L — The intervention method in this study used Phoenix dactylifera L. (dates) as the main ingredient with a standardized dose of 120 grams per day per participant, divided into three 40-gram portions over a 28-day period. The dates used were food-grade with a Certificate of Analysis (CoA) certification from a trusted supplier to ensure quality and safety of consumption. Measurement instrumentation included a digital scale with an accuracy of ±0.1 grams for daily portions, an analytical balance for high-precision measurements, and a measuring cup to ensure portion consistency. The storage and distribution system was designed using food-grade airtight containers, individual plastic bags, a cooler box for transportation, and silica gel packets for humidity control, equipped with a waterproof labeling system. Documentation and monitoring were carried out using a food diary form, a 28-day intervention calendar, and a digital camera for visual documentation.
Drug: Moringa oleifera — Moringa oleifera: The intervention method in this study used Moringa oleifera capsules as the primary therapeutic agent at a standard dose of 1000 mg per day per participant, administered in two divided doses of 500 mg each (morning and evening) for a 28-day period. The Moringa oleifera capsules used were pharmaceutical-grade capsules with appropriate quality certification from a verified supplier to ensure purity and safety for human consumption. Measurement instruments included a precision analytical balance with an accuracy of ±0.1 mg for capsule weight verification, an automatic capsule counter for dose consistency, and a calibrated measuring device to ensure uniform distribution. The storage and distribution system was implemented using pharmaceutical-grade amber glass containers to protect from light degradation, individual blister packs for daily doses, temperature-controlled storage units, and desiccant packs for humidity control, equipped with a labeling system that indicated
Other: Placebo: consumed food three times a day — consumed food three times a day: Participants received no additional intervention and only consumed food three times a day for 28 days, serving as a baseline to compare the effects of the intervention.

SUMMARY:
Postpartum depression affects 10-20% of new mothers globally, potentially disrupting breast milk production. This study aimed to provide valuable insights into effective interventions to improve the health and well-being of Postpartum Mothers with depression. This study used a randomized controlled trial design with three groups: intervention 1 (dates), intervention 2 (Moringa oleifera), and a control group. A total of 363 postpartum mothers participated, and data were collected through salivary cortisol levels (ELISA) and Beck Depression Inventory (BDI) scores to measure depression levels and breast milk production (ACIS AC-15X digital scale and Crown electric breast pump) before and after the intervention for 28 days. Data analysis was performed using paired sample t-test and the independent t-test.

ELIGIBILITY:
Eligibility Criteria:

Inclusion Criteria:

* Individuals aged 18-35 years
* Mothers with infants aged 2 weeks to 6 months
* Body Mass Index (BMI) greater than 18.7
* Scores on the Beck Depression Inventory (BDI) ranging from mild to severe depression
* Breast milk production of less than 300 g/day

Exclusion Criteria:

* Mothers with endocrine disorders
* Acute or chronic diseases
* Conditions such as hypoplastic breast tissue
* Use of combined estrogen contraceptives
* Mothers who smoke or consume alcohol

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 363 (Actual)
Dates: Start 2024-05-19 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Changes in Depression Levels of Breastfeeding Mothers (Based on BDI Scores), cortisol levels and breast milk production in each group | before the intervention and after 28 days of intervention. Assessments took place in week 1 (week 0) and week 4 (after 28 days).
  This study has more than one outcome measure with different units of measurement, so each variable should be expressed as a separate outcome measure and not combined unless a composite formula is defined. To clarify reporting, the Outcome Measures are revised as follows.
  Evaluation time points (for all outcomes): Week 0 (pre-intervention) and Week 4 (day 28 post-intervention).
  Primary/secondary outcomes (reported separately):
  1. Depression: Beck Depression Inventory (BDI) score, interval scale (unit: BDI score), measured at Week 0 and Week 4.
  2. Salivary cortisol level: Salivary cortisol concentration (unit: μg/dL), measured at Week 0 and Week 4.
  3. Breast milk production: Breast milk volume (unit: mL), measured at Week 0 and Week 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Poltekkes Kemenkes Kendari, Kendari, Southeast Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
IPD data was not provided to other researchers or outside this study because it is prohibited to share it according to the ethical approval from Poltekkes Kemenkes Kendari with number No.DP.04.03/F.XXXVI.15/004/2024 on May 6.